CLINICAL TRIAL: NCT03935958
Title: A Pilot 12 Month, Randomized, Controlled Trial of Curcumin in Kidney Transplant Recipients
Brief Title: Curcumin in Kidney Transplant Recipients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Verdure Sciences (Industry)
Responsible Party: Principal Investigator, Pierpaolo Di Cocco, Assistant Professor in Surgery, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-0321
Record Dates: First submitted 2019-04-23; First posted 2019-05-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: kidney transplantation; inflammation; vascular dysfunction; cognitive impairment; oxidative stress; graft function
MeSH Terms: conditions — Inflammation; Cognitive Dysfunction | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: 20 participants in supplement (receiving curcumin) group 20 participants in control (receiving placebo) group
  randomization 1:1
Who Masked: Participant
Masking Description: participants will not know if they are receiving curcumin or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin Arm (Arm 1) (Experimental): 20 subjects will be randomized (1:1) to this arm and receive curcumin for a year. In addition, subjects will have four study visits at Day 0, and 3, 6 and 12 months post-transplant. These study visits also include blood samples and questionnaires.
  Interventions: Dietary Supplement: Curcumin
- Placebo Arm (Arm 2) (Placebo Comparator): 20 subjects will be randomized (1:1) to this arm and receive placebo for a year. In addition, subjects will have four study visits at Day 0, and 3, 6 and 12 months post-transplant. These study visits also include blood samples and questionnaires.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — Patients will receive curcumin 2000 mg a day, for 12 months
  Other Names: Longvida
  Arms: Curcumin Arm (Arm 1)
Other: Placebo — Patients will receive placebo capsule identical in appearance and taste to the supplement, for 12 months
  Other Names: Longvida
  Arms: Placebo Arm (Arm 2)

SUMMARY:
The primary goal of this study is to investigate if curcumin is beneficial for kidney transplant recipients, a population with extensive baseline vascular dysfunction and cognitive impairment who have few treatment options. The possible mechanisms by which curcumin improves vascular function will be evaluated as well as whether curcumin improves cognitive function in these patients.

DETAILED DESCRIPTION:
Kidney transplant recipients are at increased risk of death from cardiovascular disease (CVD). Inflammation, oxidative stress and vascular dysfunction (impaired endothelial function and increased large elastic artery stiffness), are highly prevalent in kidney transplant recipients and contribute to the high incidence of CVD in this patient population. The most common cause of kidney transplant failure is interstitial fibrosis and tubular atrophy (IFTA). The incidence of IFTA is as high as 50% of kidney transplants at 1 year after transplantation. The pathophysiology of IFTA is not well understood. Possible mechanisms include chronic rejection or injury, inflammation, and drug toxicity. Kidney transplant recipients suffer from high rates of cognitive decline for which the investigators lack effective therapies. Thus, therapeutic interventions targeting inflammation, oxidative stress, vascular dysfunction, and cognitive impairment are a priority.

Curcumin may have positive effects in terms of cardiovascular and nephroprotection because of its antibacterial, antiviral, anti-inflammatory and anti-oxidative effects. The aim of this study is to elucidate the role of curcumin as a nutritional strategy to reduce cardiovascular risk factors as well as inflammation and oxidative stress in kidney transplant recipients. The study aims to examine if curcumin will improve endothelial function by reducing markers of inflammation and oxidative stress. In addition, the study will evaluate the potential benefit of curcumin on cognitive function in kidney transplant recipients.

Curcumin is a natural polyphenol with anti-inflammatory and antioxidant characteristics. Preliminary data indicate that curcumin administration improves endothelial dysfunction by reducing oxidative stress and inflammation and may improve cognitive function.

The primary goal of this study is to investigate if curcumin is beneficial for kidney transplant recipients, a population with extensive baseline vascular dysfunction and cognitive impairment who have few treatment options. The possible mechanisms by which curcumin improves vascular function will be evaluated as well as whether curcumin improves cognitive function in these patients.

Objectives:

1. Evaluate the effects of curcumin on kidney transplant graft function
2. Evaluate the effects of curcumin supplementation on cognitive function.
3. Evaluate the effects of curcumin on diabetes and cardiovascular outcomes
4. Evaluate the effects of curcumin on systemic and endothelial cell markers of inflammation and oxidative stress.

Methods:

Patients will be randomized 1:1 to receive either curcumin or placebo starting at the time of transplant or up to 2 weeks prior to transplant. Patients will be followed per standard of care for kidney transplant recipients. Additional blood (30mL) and urine samples will be drawn prior to transplant and at 3, 6 and 12 months post-transplant to be used for future analysis. There will be a total of 4 visits for this study. Additionally, two questionnaires will be distributed at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a recipient of a living donor or deceased donor kidney only transplant
2. The subject is > 18 years of age

Exclusion Criteria:

1. The subject has had a multi-organ transplant
2. Subjects that were taking curcumin pre-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Graft Outcomes | 12 months
  Change in GFR at 3, 6 and 12 months
Cognitive function & Pain | 12 months
  Change in Neuro-QOL Item Bank v2.0 at 0, 3, 6, and 12 months
Graft Outcomes | 12 months
  Difference in biopsy scores at 3 and 12 months
Cognitive function & Pain | 12 months
  Global Pain Scale at 0, 3, 6, and 12 months
Inflammation and oxidative stress | 12 months
  Markers of inflammation and oxidative stress at 0,3,6, & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Di Cocco, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali BH, Al-Salam S, Al Suleimani Y, Al Kalbani J, Al Bahlani S, Ashique M, Manoj P, Al Dhahli B, Al Abri N, Naser HT, Yasin J, Nemmar A, Al Za'abi M, Hartmann C, Schupp N. Curcumin Ameliorates Kidney Function and Oxidative Stress in Experimental Chronic Kidney Disease. Basic Clin Pharmacol Toxicol. 2018 Jan;122(1):65-73. doi: 10.1111/bcpt.12817. Epub 2017 Jul 10. PMID 28561324
- [Background] Sun X, Liu Y, Li C, Wang X, Zhu R, Liu C, Liu H, Wang L, Ma R, Fu M, Zhang D, Li Y. Recent Advances of Curcumin in the Prevention and Treatment of Renal Fibrosis. Biomed Res Int. 2017;2017:2418671. doi: 10.1155/2017/2418671. Epub 2017 May 4. PMID 28546962
- [Background] Shoskes D, Lapierre C, Cruz-Correa M, Muruve N, Rosario R, Fromkin B, Braun M, Copley J. Beneficial effects of the bioflavonoids curcumin and quercetin on early function in cadaveric renal transplantation: a randomized placebo controlled trial. Transplantation. 2005 Dec 15;80(11):1556-9. doi: 10.1097/01.tp.0000183290.64309.21. PMID 16371925